CLINICAL TRIAL: NCT03248245
Title: Improving Interprofessional Collaboration in Norwegian Primary Schools - A Cluster-randomised Study Evaluating the Effects of the LOG-model.
Brief Title: Improving Interprofessional Collaboration in Norwegian Primary Schools
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Collaborators: The Norwegian Directorate for Education and Training (Unknown)
Responsible Party: Principal Investigator, Ira Malmberg-Heimonen, Professor, Soc Sci dr., Oslo Metropolitan University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 54470 (NSD)
Record Dates: First submitted 2017-08-02; First posted 2017-08-14 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2019-08

CONDITIONS: Interprofessional Team Collaboration
Keywords: interprofessional team collaboration; primary school; learning environment; teacher's self-efficacy; teachers working ours; pupils learning outcome; cluster-randomized
MeSH Terms: interventions — Linear Models

STUDY DESIGN:
Intervention Model Description: Cluster-randomized study. After baseline, schools will be randomized to experimental and control groups schools. The LOG-model is implemented in experimental schools, while control group schools continues with their ordinary practices ("treatment as usual"). Effects on teachers are analyzed on the follow up areas: interprofessional team collaboration, teachers working hours, teacher's self-efficacy. Effects on pupils are analyzed on the follow up areas: learning environment- and outcome, early intervention. Effects on school level are analyzed on the follow up areas: special needs education, pupils learning outcome.
Who Masked: Participant
Masking Description: While the school owners, school leaders, teachers and collaborators are aware of whether their respective school have been randomized to experimental or control group, the pupils are masked for this information. They are aware that the schools participate in an intervention related to interprofessional team collaboration, but they do not know whether their school have been randomized to experimental or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LOG-model schools (Experimental): Experimental schools implement the LOG-model
  Interventions: Other: LOG-model
- Treatment as usual schools - TAU (Active Comparator): Control schools performing interprofessional team collaboration as usual
  Interventions: Other: TAU

INTERVENTIONS:
Other: LOG-model — Besides the LOG-manual, school owners and leaders receive economic compensation and the intervention team will supervise the implementation. School-owners, school leaders and teachers will participate in dialogue-seminars at the municipal level and the school level respectively. The aim is to discuss and agree on the goal and content of the work and discuss the experiences from the implementation. The main arena for discussing and practical implementation will be in local collaborating teams or "resource teams" in each school. The resource teams at schools will consist of various interprofessional competences in addition to the school leader. The main method in the LOG-model is the interchange and feedback process between the discussion of measures and the execution of these measures.
  Arms: LOG-model schools
Other: TAU — Ordinary practices related to interprofessional team collaboration
  Arms: Treatment as usual schools - TAU

SUMMARY:
This study includes designing, implementing and evaluating the effectiveness of process-based measures for improving interprofessional collaboration in Norwegian primary schools (5-7th grades). Focusing on leadership and organizational development, the overarching aim is to improve the use of existing interprofessional competence within schools. The interventions include meetings at municipal-level (strategic), school-level (operative) and class-level (operative), with feedback procedures to ensure communication between and within all levels. Also school internal and school external collaborators are involved at all levels of intervention.

In order to avoid contradictory roles, an implementation team is responsible for developing and implementing the intervention, while the research team conduct an independent evaluation. The model will be evaluated by a cluster-randomized design to evaluate the effectiveness of the intervention. The hypothesis is that schools that utilize the process-based intervention (intervention group) will improve their interprofessional team work in a way that enhances the pupil's learning- environment and teachers professional competence, self-efficacy and efficient use of working hours compared to their counterparts in the control group. We anticipate main effects to be found at pupil level, mainly through improved early assessment, intervention and efficient follow-up. The project is a collaboration between four Norwegian municipalities and includes a total of 37 Schools, half of which will be randomized to experimental condition and half to control condition.

The project is financed by The Norwegian Directorate for Education and Training with a duration of three years and three months. The project is led by Professor Ira Malmberg-Heimonen. The project is a collaboration between Faculty of Social Sciences and the Work Research Institute (AFI), at Oslo and Akerhus University College of Applied Sciences. Participants in the project are Ira Malmberg-Heimonen (project leader), Anne Grete Tøge, Therese Saltkjel, Knut Fossestøl, Elin Borg and Selma Therese Lyng. Participants in the implementation team are Øyvind Pålshaugen, Hanne Christoffersen and Christian Wittrock, also from Oslo and Akerhus University College of Applied Sciences, in addition to Torbjørn Lund from the Arctic University of Norway

DETAILED DESCRIPTION:
Comprehensive process-based intervention for improving interprofessional team collaboration in schools. A cluster-randomized study.

Start at 01.04.2017 Finnish at 30.06.2020. Funding: The Norwegian Directorate for Education and Training Collaboration: All public schools at primary level in four Norwegian municipalities

Primary schools participating in the study:

From the municipality of Ålesund: Åse, Aspøy, Blindheim, Ellingsøy, Emblem, Flisnes, Hatlane, Hessa, Larsgården, Lerstad, Spjelkavik, Vik and Stokke, and Voldsdalen.

From the municipality of Harstad: Bergseng, Bjarkøy, Harstad, Kanebogen, Kila, Lundenes, Medkila skole, Seljestad and Sørvik From the municipality of Nedre Eiker: Mjøndalen, Krokstad, Solberg, Steinberg, Stenseth and Åsen.

From the municipality of Lillehammer: Vingar, Vingrom, Søre Ål, Røyslimoen, Kringsjå, Ekrom and Buvollen (will be merged), Hammartun and Jørstadmoen

Advisory Board for the project:

Senior researcher Mary Visher, Manpower Demonstration Research Corporation (MDRC), USA Professor Nancy Cartwright, Durham University, UK, and University of California, San Diego, USA Analyst and content director Jarl Inge Wærnes, LearnLab, Oslo Norway

There are interprofessional resources in Norwegian schools and municipalities that are not fully utilized/exploited. Oslo and Akershus University College of Applied Sciences has been commissioned to design, implement and evaluate the effectiveness of a process-based model for interprofessional team collaboration in Norwegian primary schools. In order for municipal school owners and leaders to better utilize the potential related to existing interprofessional resources in schools, municipalities will implement a process-based model with a focus on leadership and better coordination of existing interprofessional resources. While the work process will be the same for all schools enrolled to experimental group, the content of the intervention will vary based on local conditions, resources and needs. A manual describes how the work process should be carried out. The model is hereafter referred to as the LOG-model, a Norwegian acronym, referring to the terms leadership, organization and coordination

The evaluation will be conducted as a cluster-randomized trial, where 37 primary schools will be randomly assigned to experimental and control groups. Schools randomized to experimental group will implement the LOG-model, while schools assign to the control group will work as previously with interprofessional collaboration. While schools in the experimental group will receive economic resources to compensate for implementing the model and participating in the research, schools randomized to control group will get, however, somewhat less financial compensation for taking part in the research. The implementation team offer supervision and support to schools randomized to the experimental group throughout the project period.

The main working method in the LOG-model is the interchange and feedback process between discursive practices, i.e. the discussion of interprofessional team collaborating measures and the execution/testing of these measures.

Staff from Oslo and Akershus College of Applied Sciences will have different roles in the project. Beside the implementation team with the role of facilitating implementation processes in schools randomized to experimental group, the process evaluation team will study implementation processes mainly based on qualitative data. The researchers in the effect-evaluation team will mainly work with quantitative data.

Prior to randomization a baseline questionnaire will be collected from the teachers and their interprofessional collaborators e.g. educational and psychological counseling services, public health nurses and child welfare social workers. Baseline information on pupils will be based on a survey data collected autumn 2017 and survey data and administrative data for follow-up + 12 and + 24 months. Long-term effects for pupils will be measured after the project has formally ended, up to 4 years after baseline, given that the Norwegian Directorate for Education and Training authorize access and deliver administrative data for follow-up.

The project will assess whether schools randomized to experimental group that are implementing the LOG-model improve their interprofessional collaboration in a way that has positive effects on learning environment, learning outcomes and early intervention for pupils. At teacher level we expect the model to increase competence for interprofessional collaboration, teacher self-efficacy and more efficient use of teachers working time.

This knowledge will inform the debate on what the effects of interprofessional team collaboration can be in schools.

The project is funded by The Norwegian Directorate for Education and Training and led by professor Ira Malmberg-Heimonen, Oslo and Akershus University College.

Participants in the project are Ira Malmberg-Heimonen (project leader), Knut Fossestøl, Øyvind Pålshagen, Elin Borg, Selma Therese Lyng, Anne Grete Tøge, Hanne Christensen, Thorbjørn Lund and Therese Saltkjel.

ELIGIBILITY:
Inclusion Criteria:

* Pupils in grades 5 - 7 in 4 municipalities and 37 primary schools
* Teachers in grades 5-7 in 4 municipalities and 37 primary schools
* Interprofessional collaborators at municipal level

Exclusion Criteria:

* NA

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4130 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Change in interprofessional team collaboration among staff | improvement from baseline (2017) to +12 (2018) months and +24 (2019) months
  Perceptions of Interprofessional Collaboration model questionnaire(teachers and collaborators)

SECONDARY OUTCOMES:
Change in teacher self-efficacy | improvement from baseline to +12 and 24 months (measured yearly)
  Norwegian teachers self-efficacy scale
Change in learning environment (teacher-level) | +12 and 24 months after baseline
  Questions from the OECD TALIS Survey (national teacher survey)
Change in teaching practices | +12 and 24 months after baseline
  Questions from the OECD TALIS Survey
Change in special needs education | change between baseline and +12 and +24 months after (measured yearly)
  amount of pupils who receive special needs education (amount at class or school level)
Change in learning enviroment (pupils) | +12 and +24 after baseline
  Questions from the Norwegian "Elevundersøkelsen" (National pupils survey)

CONTACTS AND LOCATIONS:
Locations (37):
- Norway (37):
  - Aspøy skole, Ålesund
  - Blindheim primary school, Ålesund
  - Ellingsøy primary and secondary school, Ålesund
  - Emblem skole, Ålesund
  - Flisnes skole, Ålesund
  - Hatlane skole, Ålesund
  - Hessa skole, Ålesund
  - Larsgården skole, Ålesund
  - Lerstad skole, Ålesund
  - Spjelkavik primary school, Ålesund
  - Stokke og Vik skole, Ålesund
  - Voldsdalen skole, Ålesund
  - Åse Skole, Ålesund
  - Bergseng skole, Harstad
  - Harstad skole, Harstad
  - Seljestad primary school, Harstad
  - Kanebogen skole, Harstad
  - Medkila skole, Harstad
  - Kila skole, Harstad
  - Sørvik skole, Harstad
  - Lundenes skole, Harstad
  - Bjarkøy skole, Harstad
  - Søre Ål skole, Lillehammer
  - Vingrom skole, Lillehammer
  - Vingar skole, Lillehammer
  - Hammartun skole, Lillehammer
  - Røyslimoen skole, Lillehammer
  - Kringsjå skole, Lillehammer
  - Ekrom skole, Lillehammer
  - Buvollen skole, Lillehammer
  - Jørstadmoen Skole, Lillehammer
  - Mjøndalen skole, Nedre Eiker
  - Åsen skole, Nedre Eiker
  - Steinberg Skole, Nedre Eiker
  - Krokstad skole, Nedre Eiker
  - Stenseth Skole, Nedre Eiker
  - Solberg skole, Nedre Eiker

IPD SHARING:
Plan to Share IPD: No
After embargo + 5 years after finishing study (2025)